CLINICAL TRIAL: NCT06322199
Title: Differences Between Suicide Attempters and Suicide Ideators. Influence of the Brief Therapy ASSIP on Neuropsychological Correlates and Psychological Process Factors (NePsyASSIP HT) - Project 3
Brief Title: Differences Between Suicide Attempters and Suicide Ideators. Influence of the Brief Therapy Attempted Suicide Short Intervention Program (ASSIP) on Neuropsychological Correlates and Psychological Process Factors - Project 3
Acronym: NePsyAssip HT
Status: Active, not recruiting | Type: Observational
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-02504 (Project 3)
Record Dates: First submitted 2024-03-06; First posted 2024-03-20 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Suicide, Attempted; Suicidal Ideation; Feasibility; Cost-effectiveness; Process Factors
MeSH Terms: conditions — Suicide, Attempted; Suicidal Ideation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: ASSIP (Attempted Suicide Short Intervention Program) flex — ASSIP is a specific therapy for patients after a suicide attempt. The brief therapy ASSIP consists of 3-4 sessions of approximately 50 min. each. ASSIP flex delivers ASSIP in the patient's personal environment as an outreach home treatment. The structure of the ASSIP is the same as in the regular ASSIP, but the program is delivered in the patient's environment.
  Session 1: A narrative interview is conducted, in which the patient is asked to tell her personal story, which led to the suicidal crisis. The narrative is video-recorded.
  Session 2: Using video playback of the recorded narrative, patient and therapist explore further details of the suicidal process.
  Session 3: A case conceptualization focusing on the patient's vulnerability and the trigger of the suicidal crisis is formulated in writing. A list of safety strategies for the prevention of future suicidal behavior is developed jointly with the patient.
  Regular letters are sent to patients over a period of 2 years.

SUMMARY:
The present study consists of 3 projects in total. It aims to investigate the (neuro-) psychological patterns from suicidal ideation to suicidal behavior as well as the feasibility and cost-effectiveness of ASSIP flex.

The overall aim of Project 3 is to evaluate the feasibility and cost-effectiveness of ASSIP flex over a 12-month follow-up period in terms of suicide reattempts and suicide correlates in a cohort who is attending ASSIP flex after a suicide attempt.

DETAILED DESCRIPTION:
Purpose and aims:

In project 3, the feasibility and cost-effectiveness of ASSIP flex setting over a 12-month follow-up period will be investigated. To investigate that, the present study examines the newly implemented ASSIP flex service developed and implemented at the University Hospital of Psychiatry and Psychotherapy Bern (Switzerland).

Background:

In Switzerland, approximately three people die by suicide every day, and suicide attempts exceed this number by far. As a previous suicide attempt is one of the strongest predictors of a completed suicide, it is of utmost importance to identify the people at risk. However, research has shown that traditional risk factors (e.g., depression, psychiatric disorder, etc.) reliably predict suicide ideation but poorly predict suicidal behavior. Furthermore, while effective suicide-specific interventions exist, up to 50% of the suicide attempters reject the recommended treatment, and around 60% discontinue treatment after one session. Hence, a different approach is required. In this study, three projects will be conducted. Project 3 evaluates the feasibility and cost-effectiveness of ASSIP flex.

Study design of Project 3:

The present study examines longitudinally and observationally the newly implemented ASSIP flex at the University Hospital of Psychiatry and Psychotherapy Bern (Switzerland) and four additional recruitment centers. Patients after a suicide attempt who are immobile and/or not able to participate in the regular ASSIP due to other reasons (e.g., shame or fear of stigmatization) are asked to participate in the ASSIP flex project. Moreover, the ASSIP flex will be implemented and investigated in four additional recruitment centers in Switzerland: 1) Sanatorium Kilchberg in Zurich; 2) Psychiatric Hospital, University of Zurich (PUKZH); 3) Centre Hospitalier Universitaire Vaudois (CHUV); 4) Center Neuchâtelois de Psychiatrie (CNP).

All ASSIP flex patients who have agreed to participate in Project 3 (ASSIP flex) are asked to complete a baseline assessment (filling out questionnaires) before the first ASSIP flex session. This baseline assessment is conducted in the patient's environment (i.e., where the ASSIP flex sessions are carried out).

After the baseline assessment, the participants receive ASSIP flex in their personal environment, and after each ASSIP Flex session, process measurements (therapeutic alliance) are completed. Moreover, repeated measurements are conducted after four-six weeks and 12 months follow-up to assess long-term effects.

In project 3 of this study, no randomization took place, and all participants in this group received ASSIP flex.

To investigate the feasibility and effects of ASSIP flex, therapists will also be asked to complete some questionnaires. After the last flex session of each case, they are asked to fill out a brief questionnaire to rate their experiences with this ASSIP flex case. Finally, therapists are asked one year and two years after their ASSIP training to fill out a short questionnaire about their experiences with the ASSIP flex.

ELIGIBILITY:
Inclusion Criteria:

Subjects fulfilling the following inclusion criteria are eligible for the study:

* Informed consent as documented by signature
* Age ≥ 18 years
* At least one previous suicide attempt
* Willingness to attend the ASSIP Flex

Exclusion Criteria:

The presence of any one of the following exclusion criteria will lead to exclusion of the subject:

* Serious cognitive impairment
* Any psychotic disorder
* Inability to follow the procedures of the study (e.g., insufficient mastery of the German language, previous enrolment into the current study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a past suicide attempt will be recruited at the University Hospital of Psychiatry and Psychotherapy Bern (Switzerland) and following recruitment centers:
  * Sanatorium Kilchberg Private Clinic for Psychiatry and Psychotherapy
  * Psychiatric University Hospital Zurich (PUKZH)
  * Vaud University Hospital (CHUV) in Lausanne
  * Department of General and Liaison Psychiatry CNP in Neuchâtel
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2022-09-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Suicidal ideation (Baseline, t0) | One week before the first ASSIP flex session.
  The Beck Scale for Suicide Ideation (BSI) is a clinical assessment tool designed to measure the severity of suicidal ideation in individuals. It is used in clinical and research settings to assess the risk of suicide. The BSI consists of 19 items, and each item is scored on a 3-point scale (0 to 2). The total score, which ranges from 0 to 38, reflects the severity of suicidal ideation. The minimum score is 0, indicating no suicidal ideation and the maximum score is 38, indicating the highest level of suicidal ideation. Higher scores indicate a greater severity of suicidal ideation, and thus, higher scores are generally associated with a worse outcome.
Suicidal ideation and suicidal behavior (Baseline, t0) | One week before the first ASSIP flex session.
  The Suicidal Ideation and Behavior Scale (SSEV) is a German 9-item self-report instrument. Items 1-7 assess the frequency of suicidal ideation, suicidal intention, suicidal impulses, and suicide plan (0 = never to 5 = many times every day). A total value is calculated using items 1-7, where a value of 0-30 can result. Additionally, suicide attempts during the past four weeks and the occurrence of lifetime suicide attempts are assessed with a dichotomous response format (yes/ no) and it is asked about the frequency of lifetime suicide attempts. Higher scores indicate a more severe level of suicidal ideation, which is generally associated with a worse outcome.
Suicidal ideation (Follow-up, t1) | After the three ASSIP flex sessions are completed, up to 4-6 weeks.
  The Beck Scale for Suicide Ideation (BSI) is a clinical assessment tool designed to measure the severity of suicidal ideation in individuals. It is used in clinical and research settings to assess the risk of suicide. The BSI consists of 19 items, and each item is scored on a 3-point scale (0 to 2). The total score, which ranges from 0 to 38, reflects the severity of suicidal ideation. The minimum score is 0, indicating no suicidal ideation and the maximum score is 38, indicating the highest level of suicidal ideation. Higher scores indicate a greater severity of suicidal ideation, and thus, higher scores are generally associated with a worse outcome.
Suicidal ideation and suicidal behavior (Follow-up, t1) | After the three ASSIP flex sessions are completed, up to 4-6 weeks.
  The Suicidal Ideation and Behavior Scale (SSEV) is a German 9-item self-report instrument. Items 1-7 assess the frequency of suicidal ideation, suicidal intention, suicidal impulses, and suicide plan (0 = never to 5 = many times every day). A total value is calculated using items 1-7, where a value of 0-30 can result. Additionally, suicide attempts during the past four weeks and the occurrence of lifetime suicide attempts are assessed with a dichotomous response format (yes/ no) and it is asked about the frequency of lifetime suicide attempts. Higher scores indicate a more severe level of suicidal ideation, which is generally associated with a worse outcome.
Suicidal ideation (Follow-up, t2) | 12 months after the baseline assessment.
  The Beck Scale for Suicide Ideation (BSI) is a clinical assessment tool designed to measure the severity of suicidal ideation in individuals. It is used in clinical and research settings to assess the risk of suicide. The BSI consists of 19 items, and each item is scored on a 3-point scale (0 to 2). The total score, which ranges from 0 to 38, reflects the severity of suicidal ideation. The minimum score is 0, indicating no suicidal ideation and the maximum score is 38, indicating the highest level of suicidal ideation. Higher scores indicate a greater severity of suicidal ideation, and thus, higher scores are generally associated with a worse outcome.
Suicidal ideation and suicidal behavior (Follow-up, t2) | 12 months after the baseline assessment.
  The Suicidal Ideation and Behavior Scale (SSEV) is a German 9-item self-report instrument. Items 1-7 assess the frequency of suicidal ideation, suicidal intention, suicidal impulses, and suicide plan (0 = never to 5 = many times every day). A total value is calculated using items 1-7, where a value of 0-30 can result. Additionally, suicide attempts during the past four weeks and the occurrence of lifetime suicide attempts are assessed with a dichotomous response format (yes/ no) and it is asked about the frequency of lifetime suicide attempts. Higher scores indicate a more severe level of suicidal ideation, which is generally associated with a worse outcome.

SECONDARY OUTCOMES:
Treatment costs of treatments 1 | t0) Before the first ASSIP flex session, 1 week after informed consent procedure; t1) After the intervention, 4-6 weeks after t0; t2) up to 12 months after t0
  Number of inpatient, daypatient and outpatient treatments will be assessed by DEMO.

OTHER OUTCOMES:
Sociodemographic data | t0) Before the first ASSIP flex session, 1 week after informed consent procedure; t1) After the intervention, 4-6 weeks after t0; t2) 12 months after t0
  The Sociodemographic Questionnaire (DEMO) is a 65-item questionnaire that was developed to collect sociodemographic (e.g., gender, socioeconomic status, professional status, relationship satisfaction) and health-related data (e.g., medication, inpatient and outpatient treatment).
Depressive symptoms | t0) Before the first ASSIP flex session, 1 week after informed consent procedure; t1) After the intervention, 4-6 weeks after t0; t2) 12 months after t0
  The Beck Depression Inventory (BDI-II) is a self-assessment questionnaire and contains 21 items which assess the severity of depressive symptoms. A participant's score is calculated by summing up the scores from each item. The total score ranges from 0 to 63. Values between 0 and 11 lie within the norm, between 11 and 17 moderate depressive symptoms and a total score up to 18 is assessed as a clinically relevant depressive disorder.
General sense of self-efficacy | t0) Before the first ASSIP flex session, 1 week after informed consent procedure; t1) After the intervention, 4-6 weeks after t0; t2) 12 months after t0
  The General Self-Efficacy Scale (GSE) is a 10-item self-report questionnaire to assess the general sense of self-efficacy. Items are rated from 1 (do not agree) to 4 (totally agree). The individual test score is calculated as the sum of the 10-item responses. This results in a total score of 10 to 40 points. A higher score indicates a stronger belief in one's ability to cope with and navigate different situations.
Self-Management | t0) Before the first ASSIP flex session, 1 week after informed consent procedure; t1) After the intervention, 4-6 weeks after t0; t2) 12 months after t0
  The self-management self-test (SMST) assesses self-management skills and consists of five items. The assessment is based on a five-point Likert scale (0-4 points). The items are added together so that the overall scale can have a value of 0-20 (0-4 = poor self-management, 5-8 = relatively poor self-management, 9-12 = mediocre self-management, 13-16 = fairly good self-management, 17-20 = good self-management).
Health Literacy | t0) Before the first ASSIP flex session, 1 week after informed consent procedure; t1) After the intervention, 4-6 weeks after t0; t2) 12 months after t0
  The Health Literacy Questionnaire (HLS19-Q12) assesses the general health literacy of people and contains 12 items which are assessed on a four-point Likert scale (1 = very difficult, 4 = very easy). The overall scale can have a value of 12-48. A higher score means less difficulties in accessing, understanding, evaluating and applying information to tasks related to decision-making on health topics.
Loneliness | t0) Before the first ASSIP flex session, 1 week after informed consent procedure; t1) After the intervention, 4-6 weeks after t0; t2) 12 months after t0
  The Three-Item UCLA (University of California, Los Angeles) Loneliness Scale is a short questionnaire with three items from the Revised UCLA Loneliness Scale (R-UCLA). These items can be rated from 1 (hardly ever) to 3 (often). The overall scale can have a value of 3-9. A higher score indicates a higher level of perceived loneliness. The scale is designed to measure subjective feelings of loneliness, so individuals who score higher on the UCLA Loneliness Scale report more frequent experiences of loneliness and social isolation.
Therapeutic Alliance | After the three ASSIP flex sessions are completed up to 4-6 weeks.
  The Working Alliance Inventory - short revised (WAI-SR) in German is an empirical instrument for recording the therapeutic alliance. It contains 12 items on three scales. Each item is rated on a 5-point Likert scale (rarely = 1 to always = 5). The individual test score is calculated by totaling the 12-item responses, resulting in a score between 12 and 60. A higher value means a better therapeutic alliance.
Adherence and Competence | After the three ASSIP flex sessions are completed, up to 4-6 weeks.
  Adherence and Competence Scales, elements 1-5. The ACS scales were developed using the ASSIP criteria. Therefore, five different elements were distinguished (narrative interview, video playback, case conceptualization, homework, letters). Compliance with the ASSIP manuals is ensured by means of the Adherence and Competence Scale (ACS) and its corresponding coding manual. A higher value means better adherence

CONTACTS AND LOCATIONS:
Overall Officials: Anja C. Gysin-Maillart, PD, Principal Investigator — Univerisity of Bern, University Hospital of Psychiatry, Translational Research Center; Adriana O. Frei, MSc, Study Chair — University of Bern, University Hospital of Psychiatry, Translational Research Center
Locations (4):
- Switzerland (4):
  - Centre Hospitalier universitaire vaudois (CHUV), Lausanne
  - Center Neuchâtelois de Psychiatrie, Neuchâtel
  - Psychiatric Hospital, University of Zurich (PUKZH), Zurich
  - Sanatorium Kilchberg, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peter, C. and A. Tuch, Suizidgedanken und Suizidversuche in der Schweizer Bevölkerung. Obsan Bulletin. Vol. 7. 2019, Nêuchatel. 2019.
- [Background] Bostwick JM, Pabbati C, Geske JR, McKean AJ. Suicide Attempt as a Risk Factor for Completed Suicide: Even More Lethal Than We Knew. Am J Psychiatry. 2016 Nov 1;173(11):1094-1100. doi: 10.1176/appi.ajp.2016.15070854. Epub 2016 Aug 13. PMID 27523496
- [Background] Ystgaard M, Arensman E, Hawton K, Madge N, van Heeringen K, Hewitt A, de Wilde EJ, De Leo D, Fekete S. Deliberate self-harm in adolescents: comparison between those who receive help following self-harm and those who do not. J Adolesc. 2009 Aug;32(4):875-91. doi: 10.1016/j.adolescence.2008.10.010. Epub 2008 Nov 22. PMID 19028399
- [Background] Klonsky ED, May A. Rethinking impulsivity in suicide. Suicide Life Threat Behav. 2010 Dec;40(6):612-9. doi: 10.1521/suli.2010.40.6.612. PMID 21198330
- [Background] Klonsky, E.D. and A.M. May, The three-step theory (3ST): A new theory of suicide rooted in the "ideation-to-action" framework. International Journal of Cognitive Therapy, 2015. 8(2): p. 114-129.
- [Background] May, A.M. and E.D. Klonsky, What distinguishes suicide attempters from suicide ideators? A meta-analysis of potential factors. Clinical Psychology: Science and Practice, 2016. 23(1): p. 5.
- [Background] Lizardi D, Stanley B. Treatment engagement: a neglected aspect in the psychiatric care of suicidal patients. Psychiatr Serv. 2010 Dec;61(12):1183-91. doi: 10.1176/ps.2010.61.12.1183. PMID 21123401
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Hautzinger, M., et al., Beck-depressions-inventar (BDI). Bearbeitung der deutschen Ausgabe. Testhandbuch. Bern: Huber, 1994.
- [Background] Schwarzer, R. and M. Jerusalem, Skala zur allgemeinen Selbstwirksamkeitserwartung. 1999, Berlin: Freie Universität Berlin. 2013.
- [Background] Hughes ME, Waite LJ, Hawkley LC, Cacioppo JT. A Short Scale for Measuring Loneliness in Large Surveys: Results From Two Population-Based Studies. Res Aging. 2004;26(6):655-672. doi: 10.1177/0164027504268574. PMID 18504506
- [Background] Hasler G, Klaghofer R, Buddeberg C. [The University of Rhode Island Change Assessment Scale (URICA)]. Psychother Psychosom Med Psychol. 2003 Sep-Oct;53(9-10):406-11. doi: 10.1055/s-2003-42172. German. PMID 14528410
- [Background] Gysin-Maillart, Michel, Conner, Westrin and Ehnvall (in progress).
- [Background] Munder T, Wilmers F, Leonhart R, Linster HW, Barth J. Working Alliance Inventory-Short Revised (WAI-SR): psychometric properties in outpatients and inpatients. Clin Psychol Psychother. 2010 May-Jun;17(3):231-9. doi: 10.1002/cpp.658. PMID 20013760
- [Background] Russell D, Peplau LA, Cutrona CE. The revised UCLA Loneliness Scale: concurrent and discriminant validity evidence. J Pers Soc Psychol. 1980 Sep;39(3):472-80. doi: 10.1037//0022-3514.39.3.472. PMID 7431205
- [Background] Teismann T, et al., Skala Suizidales Erleben und Verhalten (SSEV). Diagnostica. 2021; 67(3): 115-125.
- [Background] Wehmeier PM, Fox T, Doerr JM, Schnierer N, Bender M, Nater UM. Development and Validation of a Brief Measure of Self-Management Competence: The Self-Management Self-Test (SMST). Ther Innov Regul Sci. 2019 Jul 14:2168479019849879. doi: 10.1177/2168479019849879. Online ahead of print. PMID 31303020
- [Background] Beck AT, Steer RA, Ranieri WF. Scale for Suicide Ideation: psychometric properties of a self-report version. J Clin Psychol. 1988 Jul;44(4):499-505. doi: 10.1002/1097-4679(198807)44:43.0.co;2-6. PMID 3170753
- [Background] Lean M, Fornells-Ambrojo M, Milton A, Lloyd-Evans B, Harrison-Stewart B, Yesufu-Udechuku A, Kendall T, Johnson S. Self-management interventions for people with severe mental illness: systematic review and meta-analysis. Br J Psychiatry. 2019 May;214(5):260-268. doi: 10.1192/bjp.2019.54. Epub 2019 Mar 22. PMID 30898177
- [Background] Goldney RD, Fisher LJ, Wilson DH, Cheok F. Mental health literacy of those with major depression and suicidal ideation: an impediment to help seeking. Suicide Life Threat Behav. 2002 Winter;32(4):394-403. doi: 10.1521/suli.32.4.394.22343. PMID 12501964